CLINICAL TRIAL: NCT01086943
Title: Clinical Safety Study on an Eyelid Warming Device, Moist Heat Technology BLEPHASTEAM®, to Evaluate the Eyelid and Cornea Temperature in Healthy Volunteers
Brief Title: Clinical Safety Study on an Eyelid Warming Device to Evaluate the Eyelid and Cornea Temperature in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: LT2420-PI-CE-07/07
Record Dates: First submitted 2010-03-12; First posted 2010-03-15 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Eyelid Diseases
MeSH Terms: conditions — Eyelid Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- device arm (Experimental)
  Interventions: Device: LT2420

INTERVENTIONS:
Device: LT2420

SUMMARY:
The eyelid warming device is designed to relieve the symptoms of dysfunction of the glands in the eyelids.

Prospective, non comparative, open, monocentre study.

The objectives are:

* To verify and establish the temperature of the eyelids and cornea for each eye before and after 10 minutes device application
* To evaluate the ocular surface, NIBUT and IOP before and after device application
* To determine the acceptability of healthy volunteers on the practical use of this device

The subjects will attend 2 visits.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged from 18 to 80 years old.
* Healthy volunteers.
* For any contact lens wearers, they must be wearing hydrogel contact lenses (worn at least 3 times per week)
* Normal ocular examination in both eyes.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Purslow, Principal Investigator — Cardiff University
Locations (1):
- School of Optometry & Vision Sciences, Cardiff, United Kingdom